CLINICAL TRIAL: NCT00213278
Title: A Phase 2 Study of Vinblastine Sulphate Injection in Children With Recurrent or Refractory Low Grade Glioma
Brief Title: Phase 2 Study of Vinblastine in Children With Recurrent or Refractory Low Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Ontario Cancer Research Network (Network)
Responsible Party: Principal Investigator, Eric Bouffet, Section Head, Neuro-Oncology, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0020010429
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Glioma
Keywords: glioma; brain tumour; cancer; pediatrics; vinblastine sulfate
MeSH Terms: conditions — Glioma; Brain Neoplasms; Neoplasms | interventions — Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: vinblastine sulphate injection

INTERVENTIONS:
Drug: vinblastine sulphate injection — Vinblastine dose: 6 mg/m^2 (10 mg max.) route intravenous administration once a week over a period of 10 weeks. If response at week 10 is greater than or equal to stable, weekly Vinblastine will be continued for 42 weeks.

SUMMARY:
This study is examining whether Vinblastine is an effective drug to shrink low grade glioma brain tumors in children, and what the side effects are.

ELIGIBILITY:
Inclusion Criteria:

* < 21 years of age at original diagnosis
* histological verification of low grade glioma (glial tumors, neuronal tumors or chiasmatic-hypothalamic tumor) at original diagnosis
* evidence of tumor recurrence or progression by MRI or contrast CT
* Karnofsky and Lansky performance status of 0,1 or 2
* life expectancy of greater than or equal to 2 months
* adequate organ and bone marrow function within 7 days of starting treatment with Vinblastine
* absolute neutrophil count (ANC)> 1000/uL
* platelet count > 100,000/uL (transfusion independent)
* serum creatinine < 1.5 x normal for age
* written informed consent signed by subject and/or subject's parent/legal guardian

Exclusion Criteria:

* not recovered from the acute toxic effects of all prior chemotherapy, immunotherapy or radiotherapy
* chemotherapy within 2 weeks of entry in study (4 weeks if prior nitrosourea was used)
* less than 7 days since the completion of therapy with a biologic agent
* less than 2 months since cranial/spinal radiation
* receiving a stable dose of dexamethasone for less than one week

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2002-01; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To determine the response rate to Vinblastine in recurrent low grade glioma of childhood | 52 weeks

SECONDARY OUTCOMES:
To further assess the toxicity of weekly vinblastine in children treated at the currently defined maximally tolerated dose (MTD) of Vinblastine | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bouffet, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada